CLINICAL TRIAL: NCT04179513
Title: Phase I Clinical Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Multiple Doses of Gerilimzumab for Injection in Combination With Oral Methotrexate in Rheumatoid Arthritis Patients in Two Dose Groups
Brief Title: A Study to Evaluate the Safety and Tolerability of Multiple Doses of Gerilimzumab in Rheumatoid Arthritis Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Genor Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: GENOR GB224-002; V2.1
Record Dates: First submitted 2019-11-25; First posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GB224 10mg (Experimental): GB224 10mg
  Interventions: Biological: GB224 10mg
- GB224 20mg (Experimental): GB224 20mg
  Interventions: Biological: GB224 20mg

INTERVENTIONS:
Biological: GB224 10mg — 10 mg, 12subjects, abdominal subcutaneous injection, the next dose group can be initiated only after the safety and tolerability are confirmed within 4 weeks after the second dosing is given.
  Dosage and administration at enrollment are maintained (10~15 mg/week), oral administration, a total of 32 doses.
  Other Names: Methotrexate (MTX)
  Arms: GB224 10mg
Biological: GB224 20mg — 20 mg, 12subjects, abdominal subcutaneous injection, the next dose group can be initiated only after the safety and tolerability are confirmed within 4 weeks after the second dosing is given.
  Dosage and administration at enrollment are maintained (10~15 mg/week), oral administration, a total of 32 doses.
  Other Names: Methotrexate (MTX)
  Arms: GB224 20mg

SUMMARY:
The primary objective of this study is to evaluate the safety, tolerability and pharmacokinetic (PK) profiles of multiple abdominal subcutaneous injection of GB224 in combination with oral methotrexate in Chinese patients with moderate and severe active rheumatoid arthritis in two dose groups; the secondary objectives are to preliminarily evaluate the clinical efficacy such as ACR20 at week 32, ACR20, ACR50 and ACR70 at weeks 12 and 24, ACR50 and ACR70 at week 32, and DAS28 at weeks 12, 24 and 32 of multiple abdominal subcutaneous injection of GB224 in combination with oral methotrexate in Chinese patients with moderate and severe active rheumatoid arthritis in two dose groups as well as to preliminarily understand the immunogenicity and changes in pharmacodynamic variable (IL-6) of multiple abdominal subcutaneous injection of GB224 in combination with oral methotrexate in Chinese patients with moderate and severe active rheumatoid arthritis in two dose groups.

ELIGIBILITY:
Inclusion Criteria:

1. Understand the study procedures and contents, voluntarily participate in the clinical trial and sign the informed consent form;
2. Aged 18 to 75 years, males or females;
3. Subjects who have confirmed rheumatoid arthritis for at least 3 months according to 2010 American College of Rheumatology Classification Criteria (amendment);
4. The active stage is met at screening: the following 3 items should be met (based on 28 joints): swelling of 4 or more joints; tenderness of 6 or more joints; at least one of the following criteria is met: erythrocyte sedimentation rate >28mm/h or C-reactive protein >10mg/L (1.0mg/dL);
5. Subjects who have been treated with MTX treatment for at least 12 weeks before the before the use of investigational products and the dose remains stable (10~15mg/week) for at least 4 weeks;
6. The following DMARDs except MTX (including but not limited to chloroquine, hydroxychloroquine, gold preparation, penicillamine, sulfasalazine, azathioprine, cyclophosphamide, cyclosporin A, glucosinolate, auranofin etc.) are discontinued at least 4 weeks before the use of investigational products. Should any leflunomide is previously used, the subjects can be enrolled after washout with cholestyramine (8g, three times per day) for 11 days. If leflunomide is discontinued 12 weeks ago, the patients can be enrolled without washout with cholestyramine.
7. Use of TNF-α antagonists (approved orexploratory new agents) is allowed before the use of investigational products, however, it should be discontinued at least 4 weeks before administration of investigational products due to inadequate response, intolerability or economic reasons. If similar biological preparations (IL-6/IL-6R antagonists) were given before the use of investigational products, inadequate response and intolerability should be not observed and the drug should be discontinued at least 3 months ago.
8. If glucocorticoids are being administered before the use of investigational products, the dose must be stable and remains ≤10mg/d (equivalent to the dose of prednisone) for at least 4 weeks; if no glucocorticoids are used, no oral administration is given at least 4 weeks ago.
9. If the non-steroidal anti-inflammatory drugs (NSAIDs) are being administered before the use of investigational products, the dose should be stable for at least 2 weeks.
10. Female subjects of child-bearing potential have negative pregnancy test at screening; both males and females agree to adopt medically confirmed effective contraceptive measures during the entire study period and within 6 months after the end of this study.
11. Be able to understand and complete assessment forms;
12. Subjects can well communicate with the investigators and complete the study as required by the study.

Exclusion Criteria:

1. Be allergic to any exicipent of the investigational products or any other animal-derived protein, or hypersensitivity to immunoglobulin products; Subjects who are known to have medical history of allergic diseases or allergic constitution;
2. Subjects with rheumatoid arthritis with joint function classification of grade IV or subjects who combined to chair or bed;
3. Use of intramuscular injection, intravenous injection or intra-articular injection of glucocorticoids (including intramuscular injection of ACTH) within 4 weeks before the use of investigational products.
4. Inoculation with live (attenuated) vaccine within 4 weeks before the use of investigational products;
5. Treatment with interferon within 4 weeks before the use of investigational products;
6. Participation in clinical trials of other drugs within 3 months before the use of investigational products;
7. Any of the following is positive at screening: hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV-Ab), acquired immunodeficiency syndrome antibody (Anti-HIV) and anti-treponema pallidum antibody (TP-Ab);
8. Patients with known tuberculosis infection and patients with high risks for tuberculosis infection should be excluded. If patients with obsolete tuberculosis and latent tuberculosis infection (LTBI) agree to receive preventive anti-tuberculosis therapies (appendix 5) during the study period, they can be enrolled. Or, they will be excluded. (1) Known tuberculosis infection (any of the following criteria is met): active tuberculosis infection or presence of clinical signs and symptoms of suspected tuberculosis (pulmonary or extrapulmonary), presence of active tuberculosis infection involved any organ system, or symptoms of other organ systems corresponding to tuberculosis infection; (2) High risks for tuberculosis infection (any of the following criteria is met): known to be in close contact with active tuberculosis patients within 3 months before screening; subjects with low immunoligic function and with evidence showing any latent tuberculosis infection (LTBI); long stay with individuals infected with tuberculosis or long stay in medical service environment or institutions with high risks for tuberculosis transmission and infection; If patients with obsolete tuberculosis and latent tuberculosis infection (LTBI) agree to receive preventive anti-tuberculosis therapies (refer to appendix 5) during the study period and have received anti-tuberculosis monotherapy for at least 4 weeks, they can be enrolled. Or, they will be excluded. Obsolete tuberculosis: the radiology test or other imaging tests showing evidence of previous infection at screening or within the previous 3 months (obsolete tuberculosis evidence: scars of lung and/or pleural fiber; calcification of apex of lung or other sites; pulmonary hilus and /or mediastinal lymph node lesions; decreased volume of upper lobe of lung; pulmonary cavity). LTBI is defined as no evidence showing signs or symptoms of tuberculosis infection or abnormal physical examination, and chest X-ray test (other imaging tests) results showing no evidence of current tuberculosis infection, however, interferon gamma release assay (IGRA) is positive or the results of two IGRA tests are not clear.
9. Previous opportunistic infection (herpes zoster, cytomegalovirus, mycoplasma, pneumocystis carinii, histoplasma capsulatum, candida, aspergillus, mycobacterium other than mycobacterium tuberculosis etc.) within 6 months before screening;
10. Medical history of chronic infection (e.g., chronic hepatitis, chronic renal infection etc.), serious or life-threatening infection (e.g., hepatitis, pneumonitis and pyelonephritis etc.) or any current symptoms or signs indicating possible presence of infection (e.g., pyrexia, cough, urgent micturition, urodynia, abdominal pain, diarrhea, cutaneous infected wound etc.)
11. Subjects who are in high risk for infection (e.g., leg ulcer, retention catheterization, persistent or recurrent chest infection and bedridden or wheelchair-bound for a long term)
12. Medical history of lymphoproliferative disorder (including lymphoma, or signs or symptoms reflecting lymphoproliferative disorders at any time); or splenomegaly
13. Patients who previously or currently have malignant tumors within 5 years before screening (excluding adequately treated and completely cured skin basal cell carcinoma or squamous cell carcinoma, cervical in situ carcinoma);
14. Current or previous presence of congestive heart failure or medical history of congestive heart failure;
15. Current presence of interstitial lung disease or medical history of previous interstitial lung disease;
16. Current or previous presence of multiple sclerosis or other demyelinating diseases of the central nervous system or corresponding medical history of these diseases;
17. There is evidence showing that the subjects have serious, progressive and uncontrolled cardiovascular, renal, hepatic, hemopoietic, gastrointestinal, endocrine, pulmonary, nervous system disorders; and other conditions who are considered unsuitable for participating in this study at the discretion of the investigator;
18. The following abnormal laboratory variables should be excluded: white blood cells (WBC) <3.5×109/L, neutrophil count (ANC)<1.5×109/L, platelet count (PLT) <100×109/L, hemoglobin (HGB) <85g/L, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 times the upper limit of normal (ULN), alkaline phosphatase (ALP)> 2 times the upper limit of normal (ULN), serum creatinine (Cr) > 1.5 times ULN, triglycerides (TG)> 2 times ULN;
19. Subjects who currently or previously have other immune diseases (e.g., systemic lupus erythematosus, psoriasis or ankylosing spondylitis) which are considered unsuitable for participating in this study at the discretion of the investigator or subjects who have symptoms and signs of other diseases which are expected to affect the evaluation of investigational product;
20. Subjects with medical history of prosthetic joint infection and the artificial joints are still in the body;
21. Subjects who received arthroplasty for more than 3 times;
22. Subjects who received organ transplantation within 6 months before screening;
23. Lactating women;
24. Subjects who have medical history of long-term alcohol abuse or drug abuse;
25. Subjects who have insufficient communication, understanding and cooperation, or subjects who have low education level, cannot understand and correctly complete corresponding forms, subjects who have history of noncompliance with doctor's instructions to receive administration, or subjects who have other conditions which may interfere with protocol compliance of subjects (e.g., subjects who have psychiatric disorders or usually travel, and lack of motivation to participate in the study);
26. Subjects who have other diseases (e.g., clinically significant symptoms or abnormal laboratory variables) which are considered unsuitable for participating in this clinical study at the discretion of the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-08-15 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Adverse Effect, AE | Up to 224 days.
  Adverse Effect, AE
Serious Adverse Effect, SAE | Up to 224 days.
  Serious Adverse Effect, SAE
Maximum Tolerated Dose, MTD | Up to 224 days.
  Maximum Tolerated Dose, MTD
Dose Limited Toxicity, DLT | Up to 224 days.
  Dose Limited Toxicity, DLT
Cmax | Up to 224 days.
  Cmax
AUC 0-∞ | Up to 224 days.
  AUC0-∞
Accumulation Factor | Up to 224 days.
  Accumulation Factor
CL/Fsc | Up to 224 days.
  CL/Fsc
Vd/Fsc | Up to 224 days.
  Vd/Fsc
Tmax | Up to 224 days.
  Cmax, AUC0-∞, AR, CL/Fsc, Vd/Fsc, Tmax

SECONDARY OUTCOMES:
Number of patients with ACR20 | Up to 224 days.
  Number of patients with ACR20
Number of patients with ACR50 | Up to 224 days.
  Number of patients with ACR50
Number of patients with ACR70 | Up to 224 days.
  ACR70
Number of patients with DAS28 | Up to 224 days.
  Number of patients with DAS28
Anti-Drug Antibody, ADA | Up to 224 days.
  Anti-Drug Antibody, ADA
Concentration of Serum IL-6 | Up to 224 days.
  Concentration of Serum IL-6

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoguo Li, Ph.D, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No